CLINICAL TRIAL: NCT02916784
Title: Relationship Between Ability of Sit-to-stand and Types of Walking Device Used in Ambulatory Patients With Spinal Cord Injury
Brief Title: Sit-to-stand in Spinal Cord Injury Patient
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Other Study IDs: 571H104
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2015-11

CONDITIONS: Injuries, Spinal Cord
Keywords: Sit-to-stand; Walking devices
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sit-to-stand: Pass: The subjects seated on a standard armless chair with their back upright at 90 degrees against the backrest of the chair, feet placement on the floor with the heels at 10 cm behind the knees and their arms on their sides. Then they were instructed to stand up from the chair without using the arms. The ability was recorded as 'pass' if the subjects could safely rise from the chair without using their arms and with no more than contact guarding assist.
- Sit-to-stand: Fail: The subjects seated on a standard armless chair with their back upright at 90 degrees against the backrest of the chair, feet placement on the floor with the heels at 10 cm behind the knees and their arms on their sides. Then they were instructed to stand up from the chair without using the arms. The ability was recorded as 'fail' if the subjects could not rise from the chair without using their arms and/or with more than contact guarding assist.

SUMMARY:
1. Were there differences in functional ability between ambulatory individuals with SCI who passed and failed the independent sit-to-stand (iSTS) task?
2. Did the ability of iSTS relate to ability of walking as determined using a type of AAD used?
3. What were factors associated with the ability of iSTS?

DETAILED DESCRIPTION:
* To evaluate the proportion and compare functional abilities between subjects who passed and failed the independent sit-to-stand (iSTS) task.
* To assess the relationship between ability of iSTS and types of AAD used.
* To investigate factors associated with the ability of iSTS.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with iSCI from both non-traumatic and traumatic causes
* Aged at least 18 years
* Who are able to walk independently with or without AADs at least 15 meters continuously [FIM locomotor (FIM-L) scores = 5 to 7]

Exclusion Criteria:

* Any patients with conditions that might affect ambulatory ability; such as brain function disorders, visual deficits, musculoskeletal pain (VAS > 5), deformity of the musculoskeletal system, unable to follow a command of the tests, unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted in subjects with incomplete spinal cord injury (iSCI) who are able to walk independently with or without an ambulatory assistive device (AAD) from the Srinagarind hospital, KhonKaen University, Thailand.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Independent sit-to-stand test | 1 day
  Ability to perform sit-to-stand independently

SECONDARY OUTCOMES:
Lower limb support during sit-to-stand test | 1 day
  Percent of body-weight support during sit-to-stand performance
Timed up and go test | 1 day
  Ability of dynamic balance control

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya - Amatachaya, PhD, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Thailand.

IPD SHARING:
Plan to Share IPD: No